CLINICAL TRIAL: NCT05874102
Title: The Effect of Body Position on Oropharyngeal Swallow Function in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-078
Record Dates: First submitted 2023-03-28; First posted 2023-05-24 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Aspiration
MeSH Terms: interventions — URO protein, Arabidopsis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sidelying, then Upright (Active Comparator): Positioning in sidelying on radiology table for assessment, then will be positioned upright in tumbleform. Same bottle and liquid viscosities will be assessed in both positions.
  Interventions: Other: Sidelying; Other: Upright
- Upright, then Sidelying (Active Comparator): Positioned upright in tumbleform, then will be positioned sidelying on radiology table for assessment. Same bottle and liquid viscosities will be assessed in both positions.
  Interventions: Other: Sidelying; Other: Upright

INTERVENTIONS:
Other: Sidelying — Position sidelying then Upright
  Other Names: Upright
Other: Upright — Position upright then sidelying
  Other Names: Sidelying

SUMMARY:
Infants are typically fed in a cradled, upright position, however feeding specialists/SLPs often position infants in a side-lying position to promote safe, quality, and neurodevelopmentally protective feeding which is supported by currently available literature. Side-lying position is often recommended by feeding specialists to reduce the risk for aspiration and improve other components of infant swallow function. However, there is no literature directly assessing airway protection during the swallow with the infant in the side-lying versus upright positions. The goal of this study is to conduct an instrumental assessment (Modified Barium Swallow/Videofluoroscopic Swallow Study) in these different positions (upright versus side-lying) to determine if there is a difference in airway compromise. The target population are infants between post-menstrual ages of 38-56 weeks who are referred for a modified barium swallow study.

DETAILED DESCRIPTION:
Infants are typically fed in a cradled, upright position. With at-risk infants, feeding specialists may adopt a side-lying position to promote safe, quality, and neurodevelopmentally protective feeding. Current literature to support this practice suggests that side-lying position improves physiologic stability during feeding as compared to the traditional cradled or upright position. Side-lying position has several theoretical benefits based on various mechanisms including its similarity to the natural breast-feeding position, reduced hydrostatic pressure of the bottle when it is held horizontally rather than vertically above the infant, increased ease of coordinating suck-swallow-breath due to decreased flow rate, and reduced work of breathing. Another possible reason that side-lying position is beneficial is improved swallow function including decreased incidence of penetration or aspiration, which is the term for food or liquid entering the airway. Aspiration can have devastating effects on infants, particularly premature infants, including respiratory illnesses, need for increased respiratory support, inability to maintain nutrition orally, long term lung damage, and even death. Side-lying position is often recommended by feeding specialists to reduce the risk for aspiration and improve other components of infant swallow function. However, there is no literature directly assessing airway protection during the swallow with the infant in the side-lying versus upright positions.

Modified Barium Swallow Studies (MBS) are considered gold standard evaluations of swallowing function and are used to determine the safest bottle-feeding plan for medically-complex infants. MBS performed on infants typically assess multiple parameters, including suck-swallow-breathe coordination and sequencing, pharyngeal residue, timing of swallow initiation, upper esophageal sphincter opening, and presence of penetration (material entering the airway but remaining above the vocal folds) or aspiration (material entering the airway and passing below the vocal folds into the trachea). These studies have traditionally been completed in the upright/cradled position, despite the use of side-lying position clinically. However, this practice is changing, as some clinicians use side-lying during MBS to improve swallow safety and therefore inform feeding recommendations. This study aims to investigate whether there are changes in swallow function of infants fed in side-lying vs upright position during MBS. MBS will be analyzed to assess infant swallow function in side-lying position compared with swallow function in upright position. The following swallow parameters will be analyzed comparatively by position: airway invasion as defined by penetration and aspiration; location of the bolus at the time of swallow initiation, and suck-swallow-breathe coordination.

Previous literature suggests that infants fed in side-lying position are better able to control bolus rate and direction of flow than when they are fed in an upright/cradled position; however, these studies use physiologic outcomes and do not actually confirm if this hypothesized benefit is true. Pilot data found that infants were better able to protect their airway during the pharyngeal swallow, as evidenced by reduced rates of penetration or aspiration. Penetration is defined as material entering the airway during feeding but remaining above the vocal folds, whereas aspiration denotes material passing below the vocal folds towards the lungs, as measured by the Penetration-Aspiration Scale.

Side-lying position is hypothesized to reduce flow rate of liquid from the oral cavity into the pharynx, allowing the infant increased time to initiate the swallow and protect the airway. Previous literature suggests that infants fed in side-lying position are better able to control bolus rate and direction of flow than when they are fed in an upright/cradled position, leading to swallow initiation with the bolus higher in the pharyngeal cavity.

Previous research suggests that infants fed in side-lying position demonstrate improved oxygenation, which may be due to the infants' ease of coordinating breathing and swallowing during feeding. Suck-swallow-breathe coordination may be easier when fed in side-lying position because of the reduced gravitational pull of the liquid into the infant's mouth, and the increased ability to control the flow rate. Pilot data revealed that infants demonstrated fewer swallows per breath when fed in a side-lying position, which may indicate a more coordinated swallow-respiration sequence.

Pilot data revealed that airway invasion (penetration and aspiration) was statistically significantly reduced, location of the bolus at time of swallow initiation was statistically significantly higher, and number of swallows per breaths were statistically significantly lower when infants were fed in a side-lying position compared to an upright/cradled position. That pilot investigation validates the need for additional research to further define the mechanisms related to this improvement, and to determine how diagnosis and medical stability moderate these findings.

If findings support that side-lying position decreases aspiration risk, it updates the standard of care for feeding, especially for at-risk infants who are not able to undergo instrumental swallow testing. Side-lying is a no-cost strategy with the potential to enhance infant and caregiver quality of life through safe and developmentally appropriate nutritional intake. Conversely, if results indicate side-lying increases swallowing risk in certain populations, this is also significant and directs the standard of care for hospitals that routinely advise side-lying in the absence of instrumental swallow testing. This work informs best practices for clinical practitioners (e.g., SLP, RN, MD, etc.) and infant caregivers (i.e., parents) to minimize the risk of aspiration and its possible health consequences.

ELIGIBILITY:
Inclusion Criteria:

* The age of the infant at the time of the study must be between 38 to 56 weeks post-menstrual age (PMA) (American Academy of Pediatrics, 2004; Balest et al., 2021, Han et al. 2020; McGratten et al., 2020).
* Infant has been referred for an MBS by their physician based on clinical need (suspected oropharyngeal dysphagia)
* Only infants with confirmed pharyngeal dysphagia, as defined by at least one airway invasion event on their MBS, will be included in final data analysis

Exclusion Criteria:

* Infants who are deemed not medically stable enough to complete an MBS
* Infants who are deemed unable to maintain a side-lying or upright position for at least 3 minutes
* Infants who do not meet the inclusion criteria above

Ages: 38 Weeks to 56 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Airway invasion outcome | Highest rating on the Penetration-Aspiration Scale will be recorded for each trial for each infant for the entirety of the study, roughly 1 year.
  This will be measured via the Penetration-Aspiration Scale (Rosenbek et al., 1996). The PAS is an 8-point scale that is a reliable measure of airway invasion in infant bottle-feeders (Gosa & Suiter, 2011; Martin-Harris et al., 2020). The scale ranges from 1-8, with 1 indicating no airway invasion and an 8 indicating silent aspiration.

SECONDARY OUTCOMES:
Swallow initiation outcome | Lowest location of bolus (presenting highest risk) will be recorded for each trial for each infant for the entirety of the study, roughly 1 year.
  This will be measured by indicating the location of the bolus head (i.e., base of tongue-BOT, vallecula-V, pyriform sinuses-P) at the onset of base of tongue propulsion (Gosa et al., 2015).
Suck-swallow-breathe (SSwB) coordination outcome | number of sucks, swallows, and breaths will be counted for each swallowing trial for each infant for the entirety of the study, roughly 1 year.
  This will be assessed using three ratio measures: between sucks to swallows, sucks to breaths, and swallows to breaths (Barlow, 2009; Lau, 2013; Sakalidis et al., 2013; Geddes & Sakalidis, 2015). Sucks per swallows generally represents sucking efficiency, indicating how many sucks are required to form a bolus, whereas swallows to breaths is more indicative of coordination of swallow-respiration (Fucile et al., 2012, Lagarde et al., 2019; Sakalidis et al., 2013). Optimal coordination is considered a 1:1:1 SSwB ratio (Lau , 2013; Lagarde et al., 2019; Palmer, 1993).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Burnham, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No